CLINICAL TRIAL: NCT00286728
Title: Dual Diagnosis Self-Help Group Referral: Outcomes and Services Use
Brief Title: Dual Diagnosis Self-Help Referral
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 05-014
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Dual Diagnosis
Keywords: self-help groups; referral and consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Intensive referral to dual-focused self-help groups
  Interventions: Behavioral: Intensive referral to dual-focused self-help
- Arm 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Intensive referral to dual-focused self-help — 4 group sessions to introduce patients to dual focused groups
  Arms: Arm 1

SUMMARY:
This project will help counselors in substance abuse treatment programs make effective referrals of dually diagnosed patients (those with a co-occurring psychiatric disorder) to self-help groups.

DETAILED DESCRIPTION:
Background:

Dual diagnosis (psychiatric and substance use) patients' (DDPs) participation in 12-step mutual-help groups is linked to lower relapse and treatment utilization rates. However, under usual referral, many DDPs do not attend, or sustain attendance of, substance-focused groups (SFG). DDPs may benefit from dual-focused groups (DFGs).

Objectives:

(1) Implement and validate procedures to help counselors make effective referrals to DFGs. DDPs were assigned to a standard- or intensive-referral to DFG condition to determine the extent to which intensive referral, compared to standard referral, increased patients' mutual-help group participation. (2) Determine whether DDPs who received intensive referral had better substance use and psychiatric outcomes.

Methods:

DDPs entering VA outpatient mental health treatment received either standard (N=145) or intensive (N=142) referral. Standard referral consisted essentially of the counselor recommending DFG participation. The keys to intensive referral were a DFG orientation and the counselor facilitating direct contact between the patient and a DFG member, and following up on recommendations for mutual help. Patients were followed at six months (80%), one year (81%) and two years (80%) to determine whether intensive referral resulted in more DFG and SFG participation, and better substance use and psychiatric outcomes.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

* Dually diagnosed veterans entering outpatient mental health treatment

Exclusion Criteria:

* Unable to correctly answer the Orientation and Registration questions of the Mini-Mental State Examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Timko, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

REFERENCES:
- [Result] Timko C, Sutkowi A, Moos R. Patients with dual diagnoses or substance use disorders only: 12-step group participation and 1-year outcomes. Subst Use Misuse. 2010 Mar;45(4):613-27. doi: 10.3109/10826080903452421. PMID 20141467
- [Result] Timko C. Detoxification history and two-year outcomes of substance use disorder treatment and mutual-help group participation. Journal of drug issues. 2013 Jun 17; 20(10):1-18.
- [Result] Makin-Byrd K, Cronkite RC, Timko C. The influence of abuse victimization on attendance and involvement in mutual-help groups among dually diagnosed male veterans. J Subst Abuse Treat. 2011 Jul;41(1):78-87. doi: 10.1016/j.jsat.2011.02.001. Epub 2011 Mar 10. PMID 21396794
- [Result] Timko C, Cronkite RC, McKellar J, Zemore S, Moos RH. Dually diagnosed patients' benefits of mutual-help groups and the role of social anxiety. J Subst Abuse Treat. 2013 Feb;44(2):216-23. doi: 10.1016/j.jsat.2012.05.007. Epub 2012 Jul 3. PMID 22763197

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Intensive Referral: Intensive referral to dual-focused self-help groups
  Intensive referral to dual-focused self-help: 4 group sessions to introduce patients to dual focused groups
- Arm 2 Usual Care: Usual care
Period: Overall Study
Arm/Group | Arm 1 Intensive Referral | Arm 2 Usual Care
Started | 142 | 145
Completed | 106 | 116
Not Completed | 36 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Intensive Referral | Arm 2 Usual Care | Total
Number analyzed (Participants) | 142 | 145 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (9.0) | 51.2 (8.8) | 51.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 131 | 130 | 261
Region of Enrollment [Number; unit: participants]
  United States | 142 | 145 | 287

OUTCOME MEASURES:

1. Primary Outcome: Psychiatric Functioning at 6 Months
Description: Addiction Severity Index psychiatric composite ranges from 0 to 1, with 1 indicating more severe problems.
Time Frame: 6 months
Population: Explanation of Ns discrepant with patient flow: Ns with psychiatric severity scores at 6 months differ from those having completed the study at 2 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 Intensive Referral | Arm 2 Usual Care
Number analyzed (Participants) | 101 | 120
units on a scale | .333 (.199) | .387 (.228)

2. Secondary Outcome: Mental Health Services Use and Costs at 6 Months, 1 Year, and 2 Years
Time Frame: 6 months, 1 year, 2 years
Population: Access to data is no longer available.
Arm/Group | Arm 1 Intensive Referral | Arm 2 Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 Intensive Referral | Arm 2 Usual Care
Serious Adverse Events (participants affected / at risk) | 4/142 | 5/145
Other Adverse Events (participants affected / at risk) | 0/142 | 0/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Intensive Referral (N=142) | Arm 2 Usual Care (N=145)
Died (Social circumstances) | 2 | 2
Incarcerated (Social circumstances) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes